CLINICAL TRIAL: NCT05473897
Title: Head and Neck Cooling as an Emergency Department Therapy to Decrease Progression of Concussive Symptoms
Brief Title: Cooling Helmets to Decrease Concussion Symptoms
Acronym: ColdCon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit enough patients; many patients lost to follow up
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHIRB #1613
Record Dates: First submitted 2022-06-23; First posted 2022-07-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Concussion, Mild; TBI (Traumatic Brain Injury)
Keywords: Concussion; mbi; emergency medicine; catalyst cryohelmet; cooling helmet
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This research protocol will utilize a randomized controlled trial, with an interventional treatment arm and a control arm, and primary endpoints revolving around patients' post-concussion symptom severity scores. The treatment arm will receive symptomatic care (see Interventions section below) along with 30 minutes of head-neck cooling in the emergency department while being monitored for side effects. The control arm will receive symptomatic care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Catalyst Cryohelmet intervention with symptomatic care (Experimental): The treatment arm will receive symptomatic care (acetaminophen 1000mg and ondansetron 4mg) along with 30 minutes of head-neck cooling in the emergency department while being monitored for side effects.
  Interventions: Device: Catalyst Cryohelmet
- Control: symptomatic care arm (No Intervention): The control arm will receive symptomatic care (acetaminophen 1000mg and ondansetron 4mg). They will not wear any helmets.

INTERVENTIONS:
Device: Catalyst Cryohelmet — The Catalyst Cryohelmet will be used to provide head and neck cooling. It comes in three sizes based on head circumference. Once informed consent is obtained then the patient's head will be measured to provide the correct helmet size. The Cold Packs will be stored in the emergency department freezer and applied to the helmet once the helmet is ready to be applied. The Cryohelmet will be washed between uses. The Catalyst Cryohelmet is registered with the FDA as D344812. It is a Class I (minimal risk) device not requiring pre-marketing or regulatory processes.
  Arms: Catalyst Cryohelmet intervention with symptomatic care

SUMMARY:
Current therapy of Mild traumatic brain injuries (TBI) revolves around symptomatic care, rest, and return to school/sport/work after symptoms have resolved. The standard intervention for sufferers of mild traumatic brain injury is brain rest, which aims to decrease symptom intensity and duration, prevent re-injury and second impact syndrome via cessation of physical and cognitive activity, and to gradually increase activity as tolerated.

Increased brain temperature can be a secondary injury result in TBI. There are limited studies, primarily in the sports medicine literature, that show head-neck cooling can be a useful adjunct as a treatment for mild TBI. Our objective will be to evaluate concussive symptoms via the Post-Concussion Symptom Severity Score Index by conducting patient follow up interviews at different timepoints over 72 hours after an emergency department visit for the head injury where head and neck cooling was applied.

DETAILED DESCRIPTION:
There are limited studies that show head-neck cooling used as a treatment for mild TBI. Increased brain temperature can be a secondary injury result in TBI. For every degree raise in temperature, the brain's demand for oxygen and glucose increases by 6 to 10%. This elevated body temperature is associated with a worse outcome in acute brain injuries like strokes or intracerebral hemorrhages. The research hypothesize is that using head-neck cooling in the acute setting of a mild TBI may decrease the overall symptomatic period following an injury.

This research protocol will utilize a randomized controlled trial, with an interventional treatment arm and a control arm, and primary endpoints revolving around patients' post-concussion symptom severity scores. The treatment arm will receive symptomatic care (see Interventions section below) along with 30 minutes of head-neck cooling in the emergency department while being monitored for side effects. The control arm will receive symptomatic care. The main goal of this study is to evaluate if head-neck cooling of 30 minutes within the first 24 hours of a concussion will decrease the symptomatic severity index score of adults who present after a head injury. In addition, patients will receive Tylenol 500mg twice daily as well as ondansetron 4mg up to twice daily. The Catalyst Cryohelmet will be used to provide head and neck cooling. It comes in three sizes based on head circumference. Once informed consent is obtained then the patient's head will be measured to provide the correct Helmet size. The Cold Packs will be stored in the emergency department freezer and applied to the helmet once the helmet is ready to be applied. The Cryohelmet will be washed between uses. The Catalyst Cryohelmet is registered with the FDA as D344812. It is a Class I (minimal risk) device not requiring pre-marketing or regulatory processes.

Anticipated secondary outcomes include but are not limited to adverse effects relating to application of the head-neck cooling, need for further intervention in the emergency department, and return to baseline function within 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Presenting chief complaint of headache, head injury, or concussion within the first 24 hours of injury.
* Glasgow Coma Scale (GCS) > 13 on arrival.

Exclusion Criteria:

* Age < 19 years or > 65 years
* Inability to provide informed consent
* Vomiting > 2 episodes following injury
* Physical or mental disability hindering adequate response to assessment of symptoms
* Hemodynamic instability/medical condition requiring further acute life-saving medical intervention
* Known brain mass, intracranial hemorrhage, skull fracture
* Scalp abnormalities including laceration or bleeding
* Presence of ventriculoperitoneal (VP) shunt
* Known hematological malignancies, including, but not limited to: multiple myeloma, leukemia, and lymphoma
* Known history of compromised liver function, cold agglutination, cold sensitivity, cryoglobulinemia, 4
* cryofibrinogenemia, and/or a history of severe migraines
* Known contraindication to ondansetron use
* Pregnant patients

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Post-Concussion Symptom Severity Score Index case report form | 0 hour
  Initial Survey of symptoms within the first 24 hours of injury before intervention Survey Title: Case Report Form: Post-Concussion Symptom Severity Score Index Where ratings range from 0-6: 0 as no symptoms, 1-2 as mild, 2-3 moderate and 5-6 severe The following symptoms will be quantitated: headache, nausea, vomiting, balance problems, dizziness, visual problems, fatigue, sensitivity to light, sensitivity to noise, numbness or tingling, pain other than headache, feeling as if "in a fog," feeling slowed down, difficulty concentrating, difficulty remembering, drowsiness, sleeping less than usual, sleeping more than usual, trouble falling asleep, more emotional than usual, irritability, sadness, and nervousness
Post-Concussion Symptom Severity Score Index case report form | 1 hour
  Survey 1 hour after the initial survey is performed. This is approximately 30 min post-cooling helmet with medications (interventional arm) or 1hr after medications are administered (control arm).
  Survey Title: Case Report Form: Post-Concussion Symptom Severity Score Index Where ratings range from 0-6: 0 as no symptoms, 1-2 as mild, 2-3 moderate and 5-6 severe The following symptoms will be quantitated: headache, nausea, vomiting, balance problems, dizziness, visual problems, fatigue, sensitivity to light, sensitivity to noise, numbness or tingling, pain other than headache, feeling as if "in a fog," feeling slowed down, difficulty concentrating, difficulty remembering, drowsiness, sleeping less than usual, sleeping more than usual, trouble falling asleep, more emotional than usual, irritability, sadness, and nervousness
Post-Concussion Symptom Severity Score Index case report form | 48 hours
  48 hours after the injury has occurred the volunteer reports their symptoms using the Post-concussion symptom severity score index Survey Title: Case Report Form: Post-Concussion Symptom Severity Score Index Where ratings range from 0-6: 0 as no symptoms, 1-2 as mild, 2-3 moderate and 5-6 severe.
  The following symptoms will be quantitated: headache, nausea, vomiting, balance problems, dizziness, visual problems, fatigue, sensitivity to light, sensitivity to noise, numbness or tingling, pain other than headache, feeling as if "in a fog," feeling slowed down, difficulty concentrating, difficulty remembering, drowsiness, sleeping less than usual, sleeping more than usual, trouble falling asleep, more emotional than usual, irritability, sadness, and nervousness
Post-Concussion Symptom Severity Score Index case report form | 72 hours
  72 hours after the injury has occurred the volunteer reports their symptoms using the Post-concussion symptom severity score index Survey Title: Case Report Form: Post-Concussion Symptom Severity Score Index Where ratings range from 0-6: 0 as no symptoms, 1-2 as mild, 2-3 moderate and 5-6 severe The following symptoms will be quantitated: headache, nausea, vomiting, balance problems, dizziness, visual problems, fatigue, sensitivity to light, sensitivity to noise, numbness or tingling, pain other than headache, feeling as if "in a fog," feeling slowed down, difficulty concentrating, difficulty remembering, drowsiness, sleeping less than usual, sleeping more than usual, trouble falling asleep, more emotional than usual, irritability, sadness, and nervousness

SECONDARY OUTCOMES:
Adverse Effects from medication | From ED Admission to Discharge. From 1 hour up to 6 hours.
  Including development of adverse effects related to medication administration
Any other medications given during the Emergency Department (ED) stay | From ED Admission to Discharge. From 1 hour up to 6 hours.
  Any other medications besides Zofran and Tylenol given during the stay in the ED
Patient Returns to Baseline Function of 0 by 1 hour survey | 1 hour
  Scores 0 (zero) on survey questionnaire
Patient Returns to Baseline Function of 0 by 48 hour survey | 48 hours
  Scores 0 (zero) on survey questionnaire
Patient Returns to Baseline Function of 0 by 72 hour survey | 72 hours
  Scores 0 (zero) on survey questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Spectrum Health Lakeland, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
These data will not be shared with other researchers

REFERENCES:
- [Background] Vollmer BL, Kirkwood MW, Comstock RD, Currie D, Grubenhoff JA. Assessing the Clinical Utility of the Question, "Is Your Child/Are You Back to Normal?" in Pediatric Concussion Symptom Resolution. Clin Pediatr (Phila). 2018 Feb;57(2):146-151. doi: 10.1177/0009922817693300. Epub 2017 Feb 15. PMID 28198194
- [Background] Guskiewicz KM, Marshall SW, Bailes J, McCrea M, Cantu RC, Randolph C, Jordan BD. Association between recurrent concussion and late-life cognitive impairment in retired professional football players. Neurosurgery. 2005 Oct;57(4):719-26; discussion 719-26. doi: 10.1093/neurosurgery/57.4.719. PMID 16239884
- [Background] Boake C, McCauley SR, Levin HS, Pedroza C, Contant CF, Song JX, Brown SA, Goodman H, Brundage SI, Diaz-Marchan PJ. Diagnostic criteria for postconcussional syndrome after mild to moderate traumatic brain injury. J Neuropsychiatry Clin Neurosci. 2005 Summer;17(3):350-6. doi: 10.1176/jnp.17.3.350. PMID 16179657
- [Background] Gibson S, Nigrovic LE, O'Brien M, Meehan WP 3rd. The effect of recommending cognitive rest on recovery from sport-related concussion. Brain Inj. 2013;27(7-8):839-42. doi: 10.3109/02699052.2013.775494. Epub 2013 Jun 12. PMID 23758286
- [Background] Fox JL, Vu EN, Doyle-Waters M, Brubacher JR, Abu-Laban R, Hu Z. Prophylactic hypothermia for traumatic brain injury: a quantitative systematic review. CJEM. 2010 Jul;12(4):355-64. doi: 10.1017/s1481803500012471. PMID 20650030
- [Background] Sahuquillo J, Vilalta A. Cooling the injured brain: how does moderate hypothermia influence the pathophysiology of traumatic brain injury. Curr Pharm Des. 2007;13(22):2310-22. doi: 10.2174/138161207781368756. PMID 17692002
- [Background] Congeni J, Murray T, Kline P, Bouhenni R, Morgan D, Liebig C, Lesak A, McNinch NL. Preliminary Safety and Efficacy of Head and Neck Cooling Therapy After Concussion in Adolescent Athletes: A Randomized Pilot Trial. Clin J Sport Med. 2022 Jul 1;32(4):341-347. doi: 10.1097/JSM.0000000000000916. Epub 2021 Mar 10. PMID 34009790
- [Background] Gard A, Tegner Y, Bakhsheshi MF, Marklund N. Selective head-neck cooling after concussion shortens return-to-play in ice hockey players. Concussion. 2021 Apr 15;6(2):CNC90. doi: 10.2217/cnc-2021-0002. PMID 34084556
- [Background] King K, Hume PA, Hind K, Clark T. Effect of Selective Head-Neck Cooling on Signs and Symptoms of Sport Originated Brain Injury in Amateur Sports: A Pilot Study. BJSTR 21(4):16062-70